CLINICAL TRIAL: NCT06172205
Title: Infusional FOLFOX Plus Camrelizumab and Apatinib Versus HAIC-FOLFOX Plus Camrelizumab and Apatinib for Hepatocellular Carcinoma of BCLC C Stage: A Multi-center Randomized Phase III Trial
Brief Title: Infusional FOLFOX Plus Camrelizumab and Apatinib vs HAIC-FOLFOX Plus Camrelizumab and Apatinib for Advanced HCC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-984-02
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: BCLC Stage C Hepatocellular Carcinoma; Chemotherapy Effect
MeSH Terms: interventions — camrelizumab; apatinib

STUDY DESIGN:
Intervention Model Description: arm1: infusional FOLFOX plus Camrelizumab and apatinib arm2: HAIC-FOLFOX plus Camrelizumab and apatinib
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infusional FOLFOX (Experimental): Infusional mFOLFOX7 plus Camrelizumab and apatinib
  Interventions: Drug: intravenous FOLFOX7 plus Camrelizumab and apatinib
- HAIC-FOLFOX (Active Comparator): HAIC-FOLFOX plus Camrelizumab and apatinib
  Interventions: Drug: HAIC-FOLFOX plus Camrelizumab and apatinib

INTERVENTIONS:
Drug: intravenous FOLFOX7 plus Camrelizumab and apatinib — Leucovorin 200mg/m2 administered IV on Days 1 of a 21 day cycle Oxaliplatin 85 mg/m2 IV on Days 1 of a 21 day cycle Fluorouracil 5-FU continuous infusion: 400mg/m2 on D1 and then 2400mg/m2 for 46h of each 21 day cycle.
  Camrelizumab 200mg infusion on D1 for every 21 days Apatinib 250mg，po，qd for every 21 days
  Arms: Infusional FOLFOX
Drug: HAIC-FOLFOX plus Camrelizumab and apatinib — 2-h infusion of oxaliplatin at 85 mg/m2 ,a 2-3-h administration of leucovorin at 200 mg/m2 , Fluorouracil 5-FU continuous infusion: 400mg/m2 on D1 and then 2400mg/m2 for 46h. Camrelizumab (200 mg intravenously, commencing in 7 days after the first HAIC cycle and repeated every 21 days) and apatinib (250 mg daily, taken orally, beginning in 7 days after the initial HAIC cycle). Camrelizumab 200mg infusion on D1 for every 21 days Apatinib 250mg，po，qd for every 21 days.
  Arms: HAIC-FOLFOX

SUMMARY:
This is a multi-center randomized phase III clinical study of first-line intravenous FOLFOX plus Camrelizumab and apatinib versus HAIC-FOLFOX plus Camrelizumab and apatinib for BCLC C stage hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75, male or female;
2. The clinical diagnosis conforms to primary hepatocellular carcinoma (HCC) and the lesion conforms to BCLC stage C.
3. Child-pugh liver function grading: Grade A or B
4. Did not received any type of other first-line drugs such as Sorafenib
5. According to RECIST 1.1 standard, patients have at least one measurable lesion (CT/MRI scan long diameter ≥10mm or CT/MRI scan short diameter ≥15mm for lymph node lesions, and the lesion has not received radiotherapy, freezing or other local treatments);
6. ECOG PS score 0-2;
7. Expected survival ≥ 12 weeks;
8. The function of vital organs meets the following requirements (excluding the use of any blood component and cell growth factor within 14 days): Blood routine:White blood cells count ≥3.0×10^9/L Platelet count ≥70×10^9/L Hemoglobin ≥80g/L(without blood transfusion); Liver and kidney function: Serum creatinine (SCr) ≤ 1.5 times upper limit of normal value (ULN); Total bilirubin (TBIL) ≤ 3 times the upper limit of normal value (ULN); AST or ALT levels ≤ 3 times the upper limit of normal value (ULN)
9. Subjects with HBV or HCV infection should receive anti-virus treatment without interfron.
10. Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during and within six months of the end of medication;Patients with negative serum or urine pregnancy tests within 7 days prior to study inclusion and who must be non-lactating, and males should agree to use contraceptives during the study period and for 6 months after the end of the study period.
11. Patients volunteered to participate in this study and signed informed consent; Subjects have good compliance and cooperate with the follow-up.

Exclusion Criteria:

1. Have received immunotherapeutic drugs or interferon in the past.
2. Severe allergic reaction to other monoclonal antibodies, immunotherapy or chemotherapy.
3. Female subjects with pregnancy or on feeding.
4. Patients with congenital or acquired immune deficiencies.
5. Abnormal coagulation function (INR>2.0, PT>16s), have bleeding tendency or are receiving thrombolysis or anticoagulation therapy, and allow preventive use of low-dose aspirin and low-molecular-weight heparin
6. The patient has suffered from other malignant tumors at the same time (except for cured skin basal cell carcinoma and cervical carcinoma in situ)
7. The patient has active infection, fever of unknown origin within 7 days (CTCAE>2)
8. Patients with congenital or acquired immune deficiencies.
9. Severe coagulation dysfunction (INR > 2.0, PT > 16s), with a significant tendency to bleed (including but not limited to vomiting blood or passing blood in stool daily within the past 3 months);
10. Moderate to severe ascites with clinical symptoms that require therapeutic puncture or drainage, or Child-Pugh score > 2 (except for cases where imaging shows only a small amount of ascites without clinical symptoms); uncontrolled or moderate to large pleural effusion or pericardial effusion;
11. Patients are to be excluded if they have a history of gastrointestinal bleeding within 6 months prior to the start of the study treatment, or have a definite tendency for gastrointestinal bleeding, including but not limited to: bleeding-risk or severe esophageal/gastric varices, locally active ulcerative lesions, or persistently positive fecal occult blood tests.
12. Occurrence of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to the start of study treatment;
13. Occurrence of thrombotic or embolic events within 6 months prior to the start of study treatment, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction, cerebrovascular abnormalities, cerebral aneurysm), pulmonary embolism, etc.;
14. Major vascular disease within 6 months prior to the start of study treatment (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis); severe, unhealed, or dehisced wounds, as well as active ulcers or untreated fractures; Criteria for Discontinuation of Study Treatment
15. Previous or current presence of central nervous system metastases;
16. Individuals with a history of substance abuse of psychiatric medications who are unable to quit, or those with mental disorders; or those with brain metastases or hepatic encephalopathy;
17. According to the judgment of the investigator, the patients with factors that may affect the results of the study or cause the study to be terminated midway, such as alcoholism, drug abuse, other serious diseases (including mental illness) need to be treated together, severe laboratory abnormalities, accompanied by family or social factors, which will affect the safety of patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
6-mon PFSR | up to approximately 3 years
  The incidence of disease progression within the first 6 months of the patient's treatment
Hepatic Reserve Function Impairment Rate(ICG-15min) | up to approximately 3 years
  ICG-R15 is a clinical parameter that assesses the volume of remaining functional hepatocytes, which reflects the functional reserve status of the liver. It is the most commonly used indicator for measuring the severity of liver damage.

SECONDARY OUTCOMES:
mORR | up to approximately 3 years
  objective response rate based on mRECIST
ORR | up to approximately 3 years
  objective response rate based on RECISTv1.1
DOR | up to approximately 3 years
  Proportion of patients who achieved complete response (CR) or partial response (PR) at the end of treatment, based on mRECIST criteria. Patients were evaluated once every 3 cycles during the 1st to 6th treatment cycle and once every 3 months during the sequential treatment phase.
DCR | up to approximately 3 years
  The percentage of patients whose tumors shrink or stabilize for a certain period of time, including complete response (CR), partial response (PR), and stable (SD) cases. Patients were evaluated once every 3 cycles during the 1st to 6th treatment cycle and once every 3 months during the sequential treatment phase.
1y-PFSR | 1 year
  The proportion of patients who did not develop tumor progression from enrollment to 1 year of follow-up.
2y-OSR | 2 year
  Proportion of patients surviving from the start of enrollment to the full 2 years of follow-up.
OS | up to approximately 5 years
  The time between the start of treatment and the patient's death
TRAE | up to approximately 3 years
  The classification of adverse events during treatment was based on NCI-CTCAE v5.0 criteria.
conversion rate | up to approximately 3 years
  rate of unresectable converted into resectable
PFS | up to approximately 3 years
  The time from the start of treatment to the first progression of the patient's diseaseTime based on RECIST V1.1.
9-mon PFSR | up to approximately 3 years
  The incidence of disease progression within the first 9 months of the patient's treatment
18-mon OSR | 2 years
  Proportion of patients surviving from the start of enrollment to the full 18 months of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No